CLINICAL TRIAL: NCT00927927
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation, Single and Multiple Dose Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0142-0002 Administered Subcutaneously to Subjects With Rheumatoid Arthritis
Brief Title: First-in-man Trial of NNC0142-0002 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN8555-3618; 2008-008703-18 (EudraCT Number)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid | interventions — NNC0142-0002 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (15):
- SD 0.0002 mg/kg (Experimental): Subjects were injected once with NNC0142-0002 at a dose of 0.0002 mg/kg
  Interventions: Drug: NNC0142-0002
- SD 0.0012 mg/kg (Experimental): Subjects were injected once with NNC0142-0002 at a dose of 0.0012 mg/kg
  Interventions: Drug: NNC0142-0002
- SD 0.007 mg/kg (Experimental): Subjects were injected once with NNC0142-0002 at a dose of 0.007 mg/kg
  Interventions: Drug: NNC0142-0002
- SD 0.035 mg/kg (Experimental): Subjects were injected once with NNC0142-0002 at a dose of 0.035 mg/kg
  Interventions: Drug: NNC0142-0002
- SD 0.175 mg/kg (Experimental): Subjects were injected once with NNC0142-0002 at a dose of 0.175 mg/kg
  Interventions: Drug: NNC0142-0002
- SD 0.7 mg/kg (Experimental): Subjects were injected once with NNC0142-0002 at a dose of 0.7 mg/kg
  Interventions: Drug: NNC0142-0002
- SD 2.5 mg/kg (Experimental): Subjects were injected once with NNC0142-0002 at a dose of 2.5 mg/kg
  Interventions: Drug: NNC0142-0002
- SD 7.5 mg/kg (Experimental): Subjects were injected once with NNC0142-0002 at a dose of 7.5 mg/kg
  Interventions: Drug: NNC0142-0002
- SD Placebo (Experimental): Subjects were injected once with placebo
  Interventions: Drug: placebo
- MD 0.02 mg/kg (Experimental): Subjects were injected biweekly four times with NNC0142-0002 at a dose of 0.02 mg/kg
  Interventions: Drug: NNC0142-0002
- MD 0.3 mg/kg (Experimental): Subjects were injected biweekly four times with NNC0142-0002 at a dose of 0.3 mg/kg
  Interventions: Drug: NNC0142-0002
- MD 1.0 mg/kg (Experimental): Subjects were injected biweekly four times with NNC0142-0002 at a dose of 1.0 mg/kg
  Interventions: Drug: NNC0142-0002
- MD 1.6 mg/kg (Experimental): Subjects were injected biweekly four times with NNC0142-0002 at a dose of 1.6 mg/kg
  Interventions: Drug: NNC0142-0002
- MD 4.0 mg/kg (Experimental): Subjects were injected biweekly four times with NNC0142-0002 at a dose of 4.0 mg/kg
  Interventions: Drug: NNC0142-0002
- MD Placebo (Experimental): Subjects were injected biweekly four times with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0142-0002 — Single dose, ranging from 0.0002 mg/kg up to max 7.5 mg/kg, administered subcutaneously (under the skin) on day 1
  Arms: SD 0.0002 mg/kg
Drug: NNC0142-0002 — Single dose, ranging from 0.0002 mg/kg up to max 7.5 mg/kg, administered subcutaneously (under the skin) on day 1
  Arms: SD 0.0012 mg/kg
Drug: NNC0142-0002 — Single dose, ranging from 0.0002 mg/kg up to max 7.5 mg/kg, administered subcutaneously (under the skin) on day 1
  Arms: SD 0.007 mg/kg
Drug: NNC0142-0002 — Single dose, ranging from 0.0002 mg/kg up to max 7.5 mg/kg, administered subcutaneously (under the skin) on day 1
  Arms: SD 0.035 mg/kg
Drug: NNC0142-0002 — Single dose, ranging from 0.0002 mg/kg up to max 7.5 mg/kg, administered subcutaneously (under the skin) on day 1
  Arms: SD 0.175 mg/kg
Drug: NNC0142-0002 — Single dose, ranging from 0.0002 mg/kg up to max 7.5 mg/kg, administered subcutaneously (under the skin) on day 1
  Arms: SD 0.7 mg/kg
Drug: NNC0142-0002 — Single dose, ranging from 0.0002 mg/kg up to max 7.5 mg/kg, administered subcutaneously (under the skin) on day 1
  Arms: SD 2.5 mg/kg
Drug: NNC0142-0002 — Single dose, ranging from 0.0002 mg/kg up to max 7.5 mg/kg, administered subcutaneously (under the skin) on day 1
  Arms: SD 7.5 mg/kg
Drug: placebo — Single dose of 0 mg/kg administered subcutaneously (under the skin); cohort 1-7b on day 1, cohort 8-11 biweekly four times
  Arms: SD Placebo
Drug: NNC0142-0002 — Multiple dose, ranging from 0.02 mg/kg up to max 4.0 mg/kg, administered subcutaneously (under the skin) four times biweekly
  Arms: MD 0.02 mg/kg
Drug: NNC0142-0002 — Multiple dose, ranging from 0.02 mg/kg up to max 4.0 mg/kg, administered subcutaneously (under the skin) four times biweekly
  Arms: MD 0.3 mg/kg
Drug: NNC0142-0002 — Multiple dose, ranging from 0.02 mg/kg up to max 4.0 mg/kg, administered subcutaneously (under the skin) four times biweekly
  Arms: MD 1.0 mg/kg
Drug: NNC0142-0002 — Multiple dose, ranging from 0.02 mg/kg up to max 4.0 mg/kg, administered subcutaneously (under the skin) four times biweekly
  Arms: MD 1.6 mg/kg
Drug: NNC0142-0002 — Multiple dose, ranging from 0.02 mg/kg up to max 4.0 mg/kg, administered subcutaneously (under the skin) four times biweekly
  Arms: MD 4.0 mg/kg
Drug: placebo — Single dose of 0 mg/kg administered subcutaneously (under the skin); cohort 1-7b on day 1, cohort 8-11 biweekly four times
  Arms: MD Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety, tolerability, pharmacokinetic (the effect of the body on the investigated drug) and signs of clinical efficacy of increasing single doses or four repeated doses of NNC 0142-0002 in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis, characterized by a Disease Activity Score (DAS28) above 3.2, and a diagnosis of at least three months duration
* Aged between 18 and 75 years (both inclusive)
* Subjects on stable doses of methotrexate for at least 4 weeks prior to dosing
* Use of highly effective contraception during the trial (both males and females)

Exclusion Criteria:

* A chronic inflammatory autoimmune or joint disease other than RA (rheumatoid arthritis)
* An active or latent tuberculosis
* Any investigational or experimental therapy within 4 weeks or 5 half-lives (whichever is longer) prior to the screening visit
* A known significant cardio-vascular disease
* Vaccination against live virus or bacteria within 4 weeks prior to randomization
* The use of concomitant medications that are prohibited in the trial (e.g., certain DMARDs (antirheumatic therapies that are disease modifying), biologics (here: biotechnologically produced antibodies), intra-articular corticoid-injections, etc.)
* A positive test result for human immunodeficiency virus (HIV) infection, hepatitis B and/or hepatitis C, or tuberculosis skin test
* Donation of greater than or equal to 400 ml of blood within 8 weeks prior to trial entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britta Væver Bysted, DVM, PhD, Study Director — Novo Nordisk A/S
Locations (1):
- Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at one site in Germany.
Pre-assignment Details: A total of 65 subjects were randomised, but only 64 subjects were exposed to trial product. One subject withdrew consent after being randomised but before receiving any trial product.
Groups:
- SD 0.0002 mg/kg: Subjects were dosed once with NNC0142-0002 at a dose of 0.0002 mg/kg
- SD 0.0012 mg/kg: Subjects were dosed once with NNC0142-0002 at a dose of 0.0012 mg/kg
- SD 0.007 mg/kg: Subjects were dosed once with NNC0142-0002 at a dose of 0.007 mg/kg
- SD 0.035 mg/kg: Subjects were dosed once with NNC0142-0002 at a dose of 0.035 mg/kg
- SD 0.175 mg/kg: Subjects were dosed once with NNC0142-0002 at a dose of 0.175 mg/kg
- SD 0.7 mg/kg: Subjects were dosed once with NNC0142-0002 at a dose of 0.7 mg/kg
- SD 2.5 mg/kg: Subjects were dosed once with NNC0142-0002 at a dose of 2.5 mg/kg
- SD 7.5 mg/kg: Subjects were dosed once with NNC0142-0002 at a dose of 7.5 mg/kg
- SD Placebo: Subjects were dosed once with placebo
Period: Overall Study
Arm/Group | SD 0.0002 mg/kg | SD 0.0012 mg/kg | SD 0.007 mg/kg | SD 0.035 mg/kg | SD 0.175 mg/kg | SD 0.7 mg/kg | SD 2.5 mg/kg | SD 7.5 mg/kg | SD Placebo | MD 0.02 mg/kg | MD 0.3 mg/kg | MD 1.0 mg/kg | MD 1.6 mg/kg | MD 4.0 mg/kg | MD Placebo
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 5 | 6 | 5 | 5 | 9
Exposed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 5 | 5 | 5 | 5 | 9
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 8 | 3 | 5 | 4 (One subject withdrew consent after being randomised but before receiving any trial product.) | 5 | 5 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SD 0.0002 mg/kg | SD 0.0012 mg/kg | SD 0.007 mg/kg | SD 0.035 mg/kg | SD 0.175 mg/kg | SD 0.7 mg/kg | SD 2.5 mg/kg | SD 7.5 mg/kg | SD Placebo | MD 0.02 mg/kg | MD 0.3 mg/kg | MD 1.0 mg/kg | MD 1.6 mg/kg | MD 4.0 mg/kg | MD Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 5 | 5 | 5 | 5 | 9 | 64
Age, Continuous [Mean (Standard Deviation); unit: participants] | 63.0 (7.9) | 60.7 (8.1) | 66.7 (8.1) | 58.3 (5.1) | 58.7 (3.1) | 52.7 (11.0) | 49.0 (10.8) | 69.0 (4.6) | 52.8 (7.8) | 55.3 (5.0) | 56.4 (9.4) | 58.4 (5.5) | 53.0 (17.9) | 48.2 (7.7) | 53.7 (11.0) | 56.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 1 | 6 | 2 | 5 | 3 | 4 | 2 | 8 | 49
  Male | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 2 | 1 | 3 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Description: Adverse event: any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, and which does not necessarily have a causal relationship with this treatment. Serious AE: AE that at any dose level resulted in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, a congenital anomaly or birth defect, or an important medical event that may jeopardize the subject and require medical or surgical intervention.
Time Frame: Adverse events were collected for a mean (min; max) of 15.7 (6.4; 42.6) weeks for single-dose subjects, and 30.6 (12.7; 43.1) for multiple-dose subjects. Visits were scheduled until receptor occupancy was below the cut-off level for receptor positivity.
Population: All randomised subjects exposed to at least one dose of NNC0142-0002 or placebo.
Measure: Number; unit: events
Arm/Group | SD 0.0002 mg/kg | SD 0.0012 mg/kg | SD 0.007 mg/kg | SD 0.035 mg/kg | SD 0.175 mg/kg | SD 0.7 mg/kg | SD 2.5 mg/kg | SD 7.5 mg/kg | SD Placebo | MD 0.02 mg/kg | MD 0.3 mg/kg | MD 1.0 mg/kg | MD 1.6 mg/kg | MD 4.0 mg/kg | MD Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 5 | 5 | 5 | 5 | 9
events
  Adverse events | 5 | 4 | 3 | 4 | 1 | 8 | 6 | 3 | 9 | 4 | 8 | 13 | 10 | 14 | 9
  Serious AE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Concentration-time Curve (AUC)
Description: Systemic exposure to NNC0142-0002.
Time Frame: Data were collected from 0 hours to at least Day 43 (SD cohorts) and Day 85 (MD cohorts), and until the receptor occupancy was confirmed below the cut-off level for receptor positivity.
Population: All randomised subjects exposed to at least one dose of NNC0142-0002 or placebo. Serum drug concentrations after dosing with less than 0.175 mg/kg (SD cohorts) and 0.3 mg/kg (MD cohorts) were below the lower limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram×h/mL
Arm/Group | SD 0.0002 mg/kg | SD 0.0012 mg/kg | SD 0.007 mg/kg | SD 0.035 mg/kg | SD 0.175 mg/kg | SD 0.7 mg/kg | SD 2.5 mg/kg | SD 7.5 mg/kg | SD Placebo | MD 0.02 mg/kg | MD 0.3 mg/kg | MD 1.0 mg/kg | MD 1.6 mg/kg | MD 4.0 mg/kg | MD Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 5 | 5 | 5 | 5 | 9
microgram×h/mL | NA (NA) — Exposure was below lower level of quantification. | NA (NA) [NA to NA] — Exposure was below lower level of quantification. | NA (NA) [NA to NA] — Exposure was below lower level of quantification. | NA (NA) [NA to NA] — Exposure was below lower level of quantification. | 91 (306.6) [lower limit 306.6] | 4229 (12.7) [lower limit 12.7] | 16616 (35.2) [lower limit 35.2] | 87461 (29.9) [lower limit 29.9] | NA (NA) [NA to NA] — AUC was not calculated as subjects were not exposed to NNC0142-0002. | NA (NA) [NA to NA] — Exposure was below lower level of quantification. | 4034 (62.8) [lower limit 62.8] | 21883 (29.6) [lower limit 29.6] | 30212 (25.4) [lower limit 25.4] | 83307 (38.3) [lower limit 38.3] | NA (NA) [lower limit NA] — AUC was not calculated as subjects were not exposed to NNC0142-0002.

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a mean (min; max) of 15.7 (6.4; 42.6) weeks for single-dose subjects, and 30.6 (12.7; 43.1) for multiple-dose subjects. Visits were scheduled until receptor occupancy was below the cut-off level for receptor positivity.
Description: The safety analysis set included all randomised subjects exposed to at least one dose of NNC0142-0002 or placebo.
Arm/Group | SD 0.0002 mg/kg | MD 0.02 mg/kg | SD 0.0012 mg/kg | SD 0.007 mg/kg | SD 0.035 mg/kg | SD 0.175 mg/kg | SD 0.7 mg/kg | SD 2.5 mg/kg | SD 7.5 mg/kg | SD Placebo | MD 0.3 mg/kg | MD 1.0 mg/kg | MD 1.6 mg/kg | MD 4.0 mg/kg | MD Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 1/3 | 0/3 | 1/3 | 0/8 | 0/5 | 0/5 | 0/5 | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 1/3 | 3/3 | 1/3 | 3/3 | 3/3 | 1/3 | 6/8 | 4/5 | 4/5 | 5/5 | 3/5 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SD 0.0002 mg/kg (N=3) | MD 0.02 mg/kg (N=3) | SD 0.0012 mg/kg (N=3) | SD 0.007 mg/kg (N=3) | SD 0.035 mg/kg (N=3) | SD 0.175 mg/kg (N=3) | SD 0.7 mg/kg (N=3) | SD 2.5 mg/kg (N=3) | SD 7.5 mg/kg (N=3) | SD Placebo (N=8) | MD 0.3 mg/kg (N=5) | MD 1.0 mg/kg (N=5) | MD 1.6 mg/kg (N=5) | MD 4.0 mg/kg (N=5) | MD Placebo (N=9)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SD 0.0002 mg/kg (N=3) | MD 0.02 mg/kg (N=3) | SD 0.0012 mg/kg (N=3) | SD 0.007 mg/kg (N=3) | SD 0.035 mg/kg (N=3) | SD 0.175 mg/kg (N=3) | SD 0.7 mg/kg (N=3) | SD 2.5 mg/kg (N=3) | SD 7.5 mg/kg (N=3) | SD Placebo (N=8) | MD 0.3 mg/kg (N=5) | MD 1.0 mg/kg (N=5) | MD 1.6 mg/kg (N=5) | MD 4.0 mg/kg (N=5) | MD Placebo (N=9)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (5) | 3 (4) | 2 (3) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Maximum tolerated dose was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to defer data release until specified milestones, e.g. availability of a clinical trial report. Novo Nordisk reserves the right to postpone publication and/or communication for short period to protect intellectual property. Novo Nordisk reserves the right to prior review of site-specific publications and to ask for deferment of publication of individual site results until after the primary manuscript is accepted for publication.